CLINICAL TRIAL: NCT06997731
Title: Local Delivery of Hyaluronan and Minocycline as an Adjunct to Scaling and Root Planing in the Treatment of Stage 2 Grade B Periodontitis in Diabetic Patients: A Randomize Control Clinical Trial With Clinical and Microbiological Study
Brief Title: Clinical Efficacy of Local Delivery of Minocycline and Hyaluronan Gel to Treat Periodontitis in Diabetic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Enas Elgendy, Professor of oral medicine and periodontology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kafrelsheikh
Record Dates: First submitted 2025-05-12; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Periodontitis and Diabetes; Periodontitis
Keywords: minocycline gel; hyaluronan gel; periodontitis; Diabetes mellitus; microbiology; scaling and root palning
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Scaling and Root Planing with placebo gel (Placebo Comparator): Twenty sites received oral hygiene instruction and scaling& root planning with placebo gel.
  * Full mouth scaling and root planning were performed in a single visit using hand instruments (scaler and universal curette). This was followed by application of a placebo gel to each studied site.
  * Oral hygiene was performed by twice daily brushing for 2 minutes.
  Interventions: Procedure: Non -surgical treatment and oral hygiene instruction; Drug: local application of placebo gel
- Scaling& root planning followed by placement of local minocycline and Gengigel® gel (Experimental): Ten patients were treated with scaling& root planning followed by placement of local minocycline and Gengigel® gel twice weekly for 3-week 1cc for each pocket.
  Interventions: Procedure: Non -surgical treatment and oral hygiene instruction; Drug: Application of minocycline and hyaluronic acid gel.
- minocycline and Gengigel® gel without scaling and root planing (Experimental): ten patients were treated with minocycline and Gengigel® topical twice weekly for 3 week 1cc for each pocket without scaling &root planning.
  Interventions: Drug: Application of minocycline and hyaluronic acid gel.

INTERVENTIONS:
Procedure: Non -surgical treatment and oral hygiene instruction — Scaling and root planing which involves mechanical removal of sup-gingival calculus and necrotic cementum. Tis will be associated with oral hygiene instruction in the form of twice daily brushing for 2 minutes.
  Arms: Scaling and Root Planing with placebo gel; Scaling& root planning followed by placement of local minocycline and Gengigel® gel
Drug: Application of minocycline and hyaluronic acid gel. — application of minocycline and Gengigel® topical gel twice weekly for 3-week 1cc for each.
  Arms: Scaling& root planning followed by placement of local minocycline and Gengigel® gel; minocycline and Gengigel® gel without scaling and root planing
Drug: local application of placebo gel — The placebo gel will be applied in the periodontal pocket twice weekly for 3-week 1cc for each.
  Arms: Scaling and Root Planing with placebo gel

SUMMARY:
The goal of this clinical trial is to investigate the local delivery of minocycline gel 2% and 0.2% hyaluronan gel to treat periodontitis in diabetic patients as adjunctive to subgingival instrumentation. The main question it aims to answer is: Does local use of minocycline gel and hyaluronan gel as an adjunct to SRP have resulted in significant additional improvement in the clinical conditions of stage II grade B periodontitis patients when compared with SRP alone?

DETAILED DESCRIPTION:
The aim of the present study was to evaluate the clinical and microbial efficacy of local delivery of minocycline gel 2% and 0.2% hyaluronan gel (Gengigel) as an adjunctive therapy to SRP compared with SRP alone in diabetes mellitus with periodontitis patients. A total of twenty controlled diabetic patients with moderate chronic periodontitis were included in the present study. The selected patients were divided into two groups (group I and group II) and every group was divided according to the split-mouth design into applied and control side. All patients were subjected to conventional periodontal therapy (SRP) except applied side of group II. Moreover, the applied side of each group was subjected to sub gingival delivery of minocycline gel and hyaluronan gel (Gengigel) and control side was subjected to SRP, the patients followed up for three weeks. Clinical parameters used in this study included plaque index (PI), gingival index (GI), Bleeding on probing (BOP), probing pocket depth (PPD) and clinical attachment level (CAL). These parameters were measured before starting the treatment and after 3 months post treatment regimen. Sub-gingival plaque samples were taken before starting the treatment and after 1 month of treatment using sterile curette and delivered in a sterile tube containing a suitable transport media and analyzed for isolation of P. intermedia and P. gingivalis. The clinical results of both groups showed statistically significant improvement for both applied and control side which higher in applied side of group I for all clinical parameters and results of microbial evaluation showed that P. intermedia and P. gingivalis count decreased significantly after treatment in both groups especially in applied side of group I. Scaling and root planning (SRP) was effective in improving clinical and microbiological parameters in controlled diabetic patients suffering from stage II grade B periodontitis. Local use of minocycline gel and hyaluronan gel (Gengigel) as an adjunct to SRP has resulted in significant additional improvement in the clinical conditions of stage II grade B periodontitis patients when compared with SRP alone, Minocycline and hyaluronan gel (Gengigel) application results in sufficient reduction in bacterial challenge especially when combined with SRP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage II, grade B periodontitis (Attachment loss 3-4 mm and probing pocket depth ≤ 5mm) in both sides.
* Adult controlled diabetic patients (Glycosylated hemoglobin (HbA1C) in controlled diabetics ≤7%)
* Patients who can maintain good oral hygiene

Exclusion Criteria:

* History of systemic diseases other than type II diabetes
* Smoking
* Pregnant or lactating women
* Previous treatment of periodontal diseases in the last six months (People who take anti-inflammatory drugs, antibiotics, or vitamins within the previous 6 month).
* People who use mouth washes regularly ·
* Participation in other clinical trials.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth (PPD) | Probing pocket depth will be recorded at baseline and after 3 months post treatment from the gingival margines to the base of the pocket.
Clinical attachment loss (CAL) | Clinical attachment level will be recorded at baseline and 3 month post treatment.
Microbiological assessment | Porphyromonas gingivalis, Prevotella intermedia will be counted in subgingival plaque samples at baseline and after 3 months post-treatment

SECONDARY OUTCOMES:
Plaque Index (PI) | plaque index will be measured at baseline and 3 months after treatment.
Gingival index (GI) | Gingival index will be recorded at baseline and after 3 months post treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Enas Elgendy, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF